CLINICAL TRIAL: NCT01987791
Title: Comparison of Prednisone and Cyclosporine in the Treatment of Thrombocytopenia in Patients With Cirrhosis Associated With Hepatitis B in China: a Collaborative, Open-label, Real World Observational Study
Brief Title: Observation Study of Prednisone and Cyclosporine in Treatment of Thrombocytopenia in Hepatitis B Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HBV-PLT-100
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Thrombocytopenia; Hepatitis B; Cirrhosis
MeSH Terms: conditions — Thrombocytopenia; Hepatitis B; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the safety and efficacy of 12 months of low dose prednisone with low dose cyclosporine combined with entecavir in patients with thrombocytopenia associated with HBV-related cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed HBV-associated cirrhosis
* had an serum HBV DNA level of more than 500 IU per milliliter
* have compensated liver cirrhosis
* thrombocytopenia (defined as a platelet count of <30,000 per cubic millimeter)
* accompanied with bleed tendency (including petechial, episxias, ecchymosis, hemoptysis, hematemesis and hematochezia)
* have a liver-biopsy specimen indicative of cirrhosis, ultrasonography and/or computed tomographic imaging evidence of cirrhosis, or endoscopic evidence of portal hypertension(splenomegaly, ascites, and esophageal varicose)

Exclusion Criteria:

* pregnant
* hepatocellular carcinoma
* decompensated cirrhosis
* coagulation function abnormal
* had a history of other disease (e.g. aplastic anemia, autoimmune disease, idiopathic thrombocytopenia et al) that could induced thrombocytopenia
* co-infected with the human immunodeficiency virus
* co-infected with hepatitis C virus
* co-infected with hepatitis D virus
* had a coexisting serious medical or psychiatric illness
* serum creatinine level was more than 1.5 times the upper limit of the normal range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients were enrolled from 15 centers in China from January 1, 2005 to September 31, 2013.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2005-01; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
treatment failure | 12 months
  The primary efficacy outcome was treatment failure, defined as the composite of (1) any platelet count below 50×109/L after four weeks treatment; (2) significant bleeding, defined as grade 2 severity from any anatomical site as per the ITP bleeding scale that defines bleed grades (0, none; 1, mild; or 2, marked) by objective criteria of 9, based on events that occurred since the last study visit; or (3) rescue treatment administered because of severe thrombocytopenia, bleeding, or a planned invasive procedure.

SECONDARY OUTCOMES:
proportion of patients with a complete platelet count response | at 4 weeks, at 6 months , and at 12 months
  Secondary end points included proportion of patients with a complete platelet count response (platelet count of ≥ 100×109/L) without rescue treatment at 4 weeks, at 6 months , and at 12 months
proportion of patients with an overall platelet count response | at 4 weeks, at 6 months , and at 12 months
  Secondary end points included proportion of patients with an overall platelet count response (platelet count of ≥ 30×109/L with doubling from baseline) without rescue treatment at 4 weeks, at 6 months , and at 12 months